CLINICAL TRIAL: NCT01192191
Title: A Long-term Study to Evaluate the Safety and Tolerability of Fluticasone Furoate (FF)/GW642444 Inhalation Powder in Japanese Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Long-term Safety Study of Fluticasone Furoate (FF)/GW642444 in Japanese Subjects With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114156
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GW642444; COPD; Fluticasone Furoate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Furoate/GW642444 100/25mcg (Experimental): Combination inhaled corticosteroid and long-acting beta2-agonist
  Interventions: Drug: Fluticasone Furoate/GW642444 Inhalation Powder 100/25mcg
- Fluticasone Furoate/GW642444 200/25mcg (Experimental): Combination inhaled corticosteroid and long-acting beta2-agonist
  Interventions: Drug: Fluticasone Furoate/GW642444 Inhalation Powder 200/25mcg

INTERVENTIONS:
Drug: Fluticasone Furoate/GW642444 Inhalation Powder 100/25mcg — Fluticasone furoate/GW642444 inhalation powder inhaled orally once daily for 52 weeks
  Arms: Fluticasone Furoate/GW642444 100/25mcg
Drug: Fluticasone Furoate/GW642444 Inhalation Powder 200/25mcg — Fluticasone furoate/GW642444 inhalation powder inhaled orally once daily for 52 weeks
  Arms: Fluticasone Furoate/GW642444 200/25mcg

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of fluticasone furoate/GW642444 inhalation powder when administered once-daily for 52 weeks in Japanese patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Out patient at least 40 years of age
* Both genders; females childbearing potencial must be willing to use birth control method
* A diagnosis of COPD at Screening
* Subjects with a current or prior history of at least 10 pack-years of cigarett smoking at Screening
* Post-bronchodilator FEV1/FVC ratio of less than 70%
* Post-bronchodilator FEV1 of less than 80%

Exclusion Criteria:

* Current diagnosis of sthma
* Respiratory disorders other than COPD
* Upper or lower respiratory infection, or exacerbation of COPD within 4 weeka prior to Screening
* Concurrent other disease that would confound study participation or affect subject safety
* Allergies to study drugs, study drugs' excipients, medications related to study drugs
* Taking another investigational medication or medication prohibited for use during this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- Japan (20):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Toyama
  - GSK Investigational Site, Wakayama
  - GSK Investigational Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 114156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114156 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A 2-week Run-in Period was used to obtain Baseline assessment of participants. The Run-in Period was followed by a 52-week Double-blind Treatment Period and a 1-week Follow-up Period.
Groups:
- FF/VI 100/25 µg: Participants received Fluticasone Furoate (FF)/GW642444 (VI) Inhalation Powder 100/25 micrograms (µg), one puff per dose, once daily (OD) in the morning via the dry powder inhaler (DPI) for 52 weeks.
- FF/VI 200/25 µg: Participants received FF/VI Inhalation Powder 200/25 µg, one puff per dose, OD in the morning via the DPI for 52 weeks.
Period: Overall Study
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Started | 60 | 127
Completed | 49 | 106
Not Completed | 11 | 21
Not completed — Adverse Event | 7 | 12
Not completed — Participants Reached Stopping Criteria | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg | Total
Number analyzed (Participants) | 60 | 127 | 187
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.5 (7.66) | 71.0 (7.39) | 70.5 (7.49)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 11 | 13
  Male | 58 | 116 | 174
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 60 | 127 | 187

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Non-serious Adverse Event (AE) and Any Serious Adverse Event (SAE) Throughout the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury. Refer to the general AE/SAE module for a list of AEs (occurring at a frequency threshold >=5%) and SAEs.
Time Frame: From the start of investigational product to the last dose of treatment (up to Week 52/Withdrawal [WD])
Population: Intent-to-Treat (ITT) Population: all participants who had been randomized to and received at least one dose of randomized medication in the treatment period
Measure: Number; unit: Participants
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 60 | 127
Participants
  Any Non-serious AE | 36 | 93
  Any SAE | 10 | 23

2. Primary Outcome: Number of Participants With Any Drug-related AE and Any Drug-related SAE Throughout the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury. Relatedness was assessed by the investigator.
Time Frame: From the start of investigational product to the last dose of treatment (up to Week 52/Withdrawal [WD])
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 60 | 127
Participants
  Any AE | 12 | 30
  Any SAE | 1 | 2

3. Secondary Outcome: Number of Participants With Pneumonia During the Treatment Period
Description: Pneumonia is an inflammatory condition of the lung, affecting primarily the microscopic air sacs known as alveoli. All diagnoses of pneumonia (radiographically confirmed or unconfirmed) were reported as an AE or SAE. An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the ot
Time Frame: From the start of investigational product to the last dose of treatment (up to Week 52/Withdrawal [WD])
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 60 | 127
Participants
  Pneumonia recorded as an AE | 6 | 19
  Pneumonia recorded as an SAE | 4 | 9

4. Secondary Outcome: Number of Participants for the Indicated Hematological Parameters Who Experienced Low, Normal, and High Levels at Baseline (BL) and Week 52/Withdrawal (WD)
Description: Hematological parameters included: Basophils (Baso), Eosinophils (Eosin), Lymphocytes (Lymph), Monocytes (Mono), Total Neutrophils (TN), Hemoglobin (Hemo), Hematocrit (Hmcrt), Platelet Count (PT), Red Blood Cell Count (RBC Count), White Blood Cell Count (WBC Count). Data are reported as the number of participants who had low, normal, and high levels at BL (Week-2) and Week 52/WD.
Time Frame: Baseline (Week -2), and Week 52/Withdrawal (WD)
Population: ITT Population. Only participants remaining in the study and contributing evaluable data at the indicated time points were analyzed.; thus the number of participants analyzed reflects everyone in the ITT Population. The number of participants assessed for each parameter is indicated by "n=X, X".
Measure: Number; unit: Participants
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 60 | 127
Participants
  Baso, High, BL, n=60, 127 | 2 | 0
  Baso, Normal, BL, n= 60, 127 | 58 | 127
  Baso, Low, BL, n= 60, 127 | 0 | 0
  Baso, High, Week 52/WD, n=56, 122 | 1 | 1
  Baso, Normal, Week 52/WD, n=56, 122 | 55 | 121
  Baso, Low, Week 52/WD n=56, 122 | 0 | 0
  Eosin, High, BL, n=60, 127 | 5 | 15
  Eosin, Normal, BL, n=60, 127 | 55 | 112
  Eosin, Low, BL, n=60, 127 | 0 | 0
  Eosin, High, Week 52/WD, n=56, 122 | 5 | 11
  Eosin, Normal, Week 52/WD, n=56, 122 | 51 | 111
  Eosin, Low, Week 52/WD, n=56, 122 | 0 | 0
  Lymph, High, BL, n=60, 127 | 1 | 1
  Lymph, Normal, BL, n=60, 127 | 58 | 121
  Lymph, Low, BL, n=60, 127 | 1 | 5
  Lymph, High, Week 52/WD, n=56, 122 | 0 | 0
  Lymph, Normal, Week 52/WD, n=56, 122 | 51 | 108
  Lymph, Low, Week 52/WD, n=56, 122 | 5 | 14
  Mono, High, BL, n=60, 127 | 9 | 8
  Mono, Normal, BL, n=60, 127 | 51 | 119
  Mono, Low, BL, n=60, 127 | 0 | 0
  Mono, High, Week 52/WD, n=56, 122 | 7 | 14
  Mono, Normal, Week 52/WD, n=56, 122 | 49 | 108
  Mono, Low, Week 52/WD, n=56, 122 | 0 | 0
  TN, High, BL, n=60, 127 | 0 | 5
  TN, Normal, BL, n=60, 127 | 58 | 119
  TN, Low, BL, n=60, 127 | 2 | 3
  TN, High, Week 52/WD, n=56, 122 | 4 | 11
  TN, Normal, Week 52/WD, n=56, 122 | 52 | 111
  TN, Low, Week 52/WD, n=56, 122 | 0 | 0
  Hemo, High, BL, n=60, 127 | 1 | 2
  Hemo, Normal, BL, n=60, 127 | 48 | 112
  Hemo, Low, BL, n=60, 127 | 11 | 13
  Hemo, High, Week 52/WD, n=56, 122 | 0 | 0
  Hemo, Normal, Week 52/WD, n=56, 122 | 45 | 108
  Hemo, Low, Week 52/WD, n=56, 122 | 11 | 14
  Hmcrt, High, BL, n=60, 127 | 4 | 13
  Hmcrt, Normal, BL, n=60, 127 | 50 | 110
  Hmcrt, Low, BL, n=60, 127 | 6 | 4
  Hmcrt, High, Week 52/WD, n=56, 122 | 1 | 8
  Hmcrt, Normal, Week 52/WD, n=56, 122 | 50 | 106
  Hmcrt, Low, Week 52/WD, n=56, 122 | 5 | 8
  PT, High, BL, n=60, 127 | 1 | 0
  PT, Normal, BL, n=60, 127 | 57 | 124
  PT, Low, BL, n=60, 127 | 2 | 3
  PT, High, Week 52/WD, n=56, 122 | 2 | 4
  PT, Normal, Week 52/WD, n=56, 122 | 51 | 116
  PT, Low, Week 52/WD, n=56, 122 | 3 | 2
  RBC Count, High, BL, n=60, 127 | 0 | 4
  RBC Count, Normal, BL, n=60, 127 | 53 | 111
  RBC Count, Low, BL, n=60, 127 | 7 | 12
  RBC Count, High, Week 52/WD, n=56, 122 | 0 | 2
  RBC Count, Normal, Week 52/WD, n=56, 122 | 47 | 107
  RBC Count, Low, Week 52/WD, n=56, 122 | 9 | 13
  WBC Count, High, BL, n=60, 127 | 2 | 6
  WBC Count, Normal, BL, n=60, 127 | 57 | 119
  WBC Count, Low, BL, n=60, 127 | 1 | 2
  WBC Count, High, Week 52/WD, n=56, 122 | 3 | 4
  WBC Count, Normal, Week 52/WD, n=56, 122 | 52 | 116
  WBC Count, Low, Week 52/WD, n=56, 122 | 1 | 2

5. Secondary Outcome: Number of Participants for the Indicated Clinical Chemistry and Urinalysis Parameters Who Experienced a Low, Normal, and High Levels at Baseline (BL) and Week 52/Withdrawal (WD)
Description: Clinical chemistry and urinalysis parameters included: Albumin, Alkaline Phosphatase (AP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Bilirubin (Direct [BD], Indirect [BI], and Total [BT]), Creatine Kinase (CK), Chloride, Carbon Dioxide content/Bicarbonate (CO2/BC), Creatinine, Gamma Glutamyl Transferase (GGT), Glucose, Potassium, Lactate Dehydrogenase (LDH), Sodium, Urine pH, Urine Specific Gravity (USG),Total Protein (TP), Urea/Blood urea nitrogen (BUN), and Uric Acid (UA). Data are reported as the number of participants who had low, normal, and high levels at BL (Week-2) and Week 52/WD.
Time Frame: Baseline (Week -2), and Week 52/Withdrawal (WD
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 60 | 127
Participants
  Albumin, High, BL, n=60, 127 | 0 | 2
  Albumin, Normal, BL, n=60, 127 | 56 | 112
  Albumin, Low, BL, n=60, 127 | 4 | 13
  Albumin, High, Week 52/WD, n=56, 122 | 0 | 1
  Albumin, Normal, Week 52/WD, n=56, 122 | 49 | 99
  Albumin, Low, Week 52/WD, n=56, 122 | 7 | 22
  AP, High, BL, n=60, 127 | 4 | 10
  AP, Normal, BL, n=60, 127 | 56 | 117
  AP, Low, BL, n=60, 127 | 0 | 0
  AP, High, Week 52/WD, n=56, 122 | 5 | 6
  AP, Normal, Week 52/WD, n=56, 122 | 51 | 116
  AP, Low, Week 52/WD, n=56, 122 | 0 | 0
  ALT, High, BL, n=60, 127 | 4 | 9
  ALT, Normal, BL, n=60, 127 | 56 | 117
  ALT, Low, BL, n=60, 127 | 0 | 1
  ALT, High, Week 52/WD, n=56, 122 | 4 | 6
  ALT, Normal, Week 52/WD, n=56, 122 | 52 | 116
  ALT, Low, Week 52/WD, n=56, 122 | 0 | 0
  AST, High, BL, n=60, 127 | 5 | 11
  AST, Normal, BL, n=60, 127 | 55 | 116
  AST, Low, BL, n=60, 127 | 0 | 0
  AST, High, Week 52/WD, n=56, 122 | 3 | 5
  AST, Normal, Week 52/WD, n=56, 122 | 53 | 117
  AST, Low, Week 52/WD, n=56, 122 | 0 | 0
  BD, High, BL, n=60, 127 | 7 | 4
  BD, Normal, BL, n=60, 127 | 53 | 123
  BD, Low, BL, n=60, 127 | 0 | 0
  BD, High, Week 52/WD, n=56, 122 | 3 | 4
  BD, Normal, Week 52/WD, n=56, 122 | 53 | 118
  BD, Low, Week 52/WD, n=56, 122 | 0 | 0
  BI, High, BL, n=60, 127 | 4 | 1
  BI, Normal, BL, n=60, 127 | 56 | 126
  BI, Low, BL, n=60, 127 | 0 | 0
  BI, High, Week 52/WD, n=56, 122 | 3 | 2
  BI, Normal, Week 52/WD, n=56, 122 | 53 | 120
  BI, Low, Week 52/WD, n=56, 122 | 0 | 0
  BT, High, BL, n=60, 127 | 6 | 5
  BT, Normal, BL, n=60, 127 | 54 | 122
  BT, Low, BL, n=60, 127 | 0 | 0
  BT, High, Week 52/WD, n=56, 122 | 6 | 3
  BT, Normal, Week 52/WD, n=56, 122 | 50 | 119
  BT, Low, Week 52/WD, n=56, 122 | 0 | 0
  CK, High, BL, n=60, 127 | 6 | 10
  CK, Normal, BL, n=60, 127 | 48 | 102
  CK, Low, BL, n=60, 127 | 6 | 15
  CK, High, Week 52/WD, n=56, 122 | 7 | 7
  CK, Normal, Week 52/WD, n=56, 122 | 44 | 92
  CK, Low, Week 52/WD, n=56, 122 | 5 | 23
  Chloride, High, BL, n=60, 127 | 1 | 0
  Chloride, Normal, BL, n=60, 127 | 58 | 124
  Chloride, Low, BL, n=60, 127 | 1 | 3
  Chloride, High, Week 52/WD, n=56, 122 | 2 | 6
  Chloride, Normal, Week 52/WD, n=56, 122 | 54 | 115
  Chloride, Low, Week 52/WD, n=56, 122 | 0 | 1
  CO2/BC, High, BL, n=60, 127 | 0 | 1
  CO2/BC, Normal, BL, n=60, 127 | 57 | 120
  CO2/BC, Low, BL, n=60, 127 | 3 | 6
  CO2/BC, High, Week 52/WD, n=56, 121 | 0 | 1
  CO2/BC, Normal, Week 52/WD, n=56, 121 | 48 | 116
  CO2/BC, Low, Week 52/WD, n=56, 121 | 8 | 4
  Creatinine, High, BL, n=60, 127 | 8 | 9
  Creatinine, Normal, BL, n=60, 127 | 50 | 115
  Creatinine, Low, BL, n=60, 127 | 2 | 3
  Creatinine, High, Week 52/WD, n=56, 122 | 6 | 10
  Creatinine, Normal, Week 52/WD, n=56, 122 | 47 | 108
  Creatinine, Low, Week 52/WD, n=56, 122 | 3 | 4
  GGT, High, BL, n=60, 127 | 9 | 25
  GGT, Normal, BL, n=60, 127 | 51 | 102
  GGT, Low, BL, n=60, 127 | 0 | 0
  GGT, High, Week 52/WD, n=56, 122 | 10 | 19
  GGT, Normal, Week 52/WD, n=56, 122 | 46 | 103
  GGT, Low, Week 52/WD, n=56, 122 | 0 | 0
  Glucose, High, BL, n=60, 127 | 16 | 58
  Glucose, Normal, BL, n=60, 127 | 43 | 65
  Glucose, Low, BL, n=60, 127 | 1 | 4
  Glucose, High, Week 52/WD, n=56, 122 | 26 | 56
  Glucose, Normal, Week 52/WD, n=56, 122 | 30 | 65
  Glucose, Low, Week 52/WD, n=56, 122 | 0 | 1
  Potassium, High, BL, n=60, 127 | 2 | 5
  Potassium, Normal, BL, n=60, 127 | 54 | 116
  Potassium, Low, BL, n=60, 127 | 4 | 6
  Potassium, High, Week 52/WD, n=56, 122 | 1 | 5
  Potassium, Normal, Week 52/WD, n=56, 122 | 53 | 111
  Potassium, Low, Week 52/WD, n=56, 122 | 2 | 6
  LDH, High, BL, n=60, 127 | 1 | 9
  LDH, Normal, BL, n=60, 127 | 59 | 116
  LDH, Low, BL, n=60, 127 | 0 | 2
  LDH, High, Week 52/WD, n=56, 122 | 4 | 10
  LDH, Normal, Week 52/WD, n=56, 122 | 52 | 111
  LDH, Low, Week 52/WD, n=56, 122 | 0 | 1
  Sodium, High, BL, n=60, 127 | 0 | 0
  Sodium, Normal, BL, n=60, 127 | 58 | 125
  Sodium, Low, BL, n=60, 127 | 2 | 2
  Sodium, High, Week 52/WD, n=56, 122 | 0 | 0
  Sodium, Normal, Week 52/WD, n=56, 122 | 55 | 120
  Sodium, Low, Week 52/WD, n=56, 122 | 1 | 2
  Urine pH, High, BL, n=60, 127 | 0 | 1
  Urine pH, Normal, BL, n=60, 127 | 60 | 126
  Urine pH, Low, BL, n=60, 127 | 0 | 0
  Urine pH, High, Week 52/WD, n=56, 122 | 0 | 0
  Urine pH, Normal, Week 52/WD, n=56, 122 | 56 | 122
  Urine pH, Low, Week 52/WD, n=56, 122 | 0 | 0
  USG, High, BL, n=60, 127 | 2 | 1
  USG, Normal, BL, n=60, 127 | 58 | 126
  USG, Low, BL, n=60, 127 | 0 | 0
  USG, High, Week 52/WD, n=56, 122 | 2 | 0
  USG, Normal, Week 52/WD, n=56, 122 | 54 | 122
  USG, Low, Week 52/WD, n=56, 122 | 0 | 0
  TP, High, BL, n=60, 127 | 1 | 3
  TP, Normal, BL, n=60, 127 | 55 | 118
  TP, Low, BL, n=60, 127 | 4 | 6
  TP, High, Week 52/WD, n=56, 122 | 1 | 3
  TP, Normal, Week 52/WD, n=56, 122 | 49 | 102
  TP, Low, Week 52/WD, n=56, 122 | 6 | 17
  Urea/BUN, High, BL, n=60, 127 | 5 | 13
  Urea/BUN, Normal, BL, n=60, 127 | 54 | 114
  Urea/BUN, Low, BL, n=60, 127 | 1 | 0
  Urea/BUN, High, Week 52/WD, n=56, 122 | 8 | 5
  Urea/BUN, Normal, Week 52/WD, n=56, 122 | 48 | 116
  Urea/BUN, Low, Week 52/WD, n=56, 122 | 0 | 1
  UA, High, BL, n=60, 127 | 13 | 22
  UA, Normal, BL, n=60, 127 | 46 | 102
  UA, Low, BL, n=60, 127 | 1 | 3
  UA, High, Week 52/WD, n=56, 122 | 13 | 23
  UA, Normal, Week 52/WD, n=56, 122 | 42 | 92
  UA, Low, Week 52/WD, n=56, 122 | 1 | 7

6. Secondary Outcome: Number of Participants for the Indicated Urinalysis Parameters Tested by Dipstick at Baseline (BL) and Week 52/Withdrawal (WD)
Description: Urinalysis parameters included: Urine Occult Blood (UOB), Urine Glucose (UG), Urine Ketones (UK), Urine Protein (UP), and Urine Leukocyte Esterase test for detecting White Blood Cell (UWBC). The dipstick was a strip used to detect the presence or absence of these parameters in the urine sample. The dipstick test gives results in a semi-quantitative manner, and results can be read as negative (Neg), Trace, 1+, 2+, and 3+, indicating proportional concentrations in the urine sample. Data are reported as the number of participants who had neg, trace, 1+, 2+, and 3+ levels at Baseline (Week -2) and Week 52/WD.
Time Frame: Baseline (Week -2), Week 52/Withdrawal (WD)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 60 | 127
Participants
  UOB, Neg, BL, n=60, 127 | 54 | 112
  UOB, Trace, BL, n=60, 127 | 4 | 6
  UOB, 1+, BL, n=60, 127 | 1 | 5
  UOB, 2+, BL, n=60, 127 | 1 | 2
  UOB, 3+, BL, n=60, 127 | 0 | 2
  UOB, Neg, Week 52/WD, n=56, 122 | 51 | 103
  UOB, Trace, Week 52/WD, n=56, 122 | 3 | 11
  UOB, 1+, Week 52/WD, n=56, 122 | 1 | 5
  UOB, 2+, Week 52/WD, n=56, 122 | 1 | 1
  UOB, 3+, Week 52/WD, n=56, 122 | 0 | 2
  UG, Neg, BL, n=60, 127 | 54 | 117
  UG, Trace, BL, n=60, 127 | 3 | 4
  UG, 1+, BL, n=60, 127 | 2 | 1
  UG, 2+, BL, n=60, 127 | 1 | 2
  UG, 3+, BL, n=60, 127 | 0 | 3
  UG, Neg, Week 52/WD, n=56, 122 | 49 | 109
  UG, Trace, Week 52/WD, n=56, 122 | 2 | 5
  UG, 1+, Week 52/WD, n=56, 122 | 3 | 1
  UG, 2+, Week 52/WD, n=56, 122 | 2 | 5
  UG, 3+, Week 52/WD, n=56, 122 | 0 | 2
  UK, Neg, BL, n=60, 127 | 60 | 127
  UK, Trace, BL, n=60, 127 | 0 | 0
  UK, 1+, BL, n=60, 127 | 0 | 0
  UK, 2+, BL, n=60, 127 | 0 | 0
  UK, 3+, BL, n=60, 127 | 0 | 0
  UK, Neg, Week 52/WD, n=56, 122 | 56 | 122
  UK, Trace, Week 52/WD, n=56, 122 | 0 | 0
  UK, 1+, Week 52/WD, n=56, 122 | 0 | 0
  UK, 2+, Week 52/WD, n=56, 122 | 0 | 0
  UK, 3+, Week 52/WD, n=56, 122 | 0 | 0
  UP, Neg, BL, n=60, 127 | 48 | 103
  UP, Trace, BL, n=60, 127 | 10 | 13
  UP, 1+, BL, n=60, 127 | 2 | 8
  UP, 2+, BL, n=60, 127 | 0 | 3
  UP, 3+, BL, n=60, 127 | 0 | 0
  UP, Neg, Week 52/WD, n=56, 122 | 41 | 92
  UP, Trace, Week 52/WD, n=56, 122 | 10 | 20
  UP, 1+, Week 52/WD, n=56, 122 | 4 | 8
  UP, 2+, Week 52/WD, n=56, 122 | 1 | 2
  UP, 3+, Week 52/WD, n=56, 122 | 0 | 0
  UWBC, Neg, BL, n=60, 127 | 58 | 120
  UWBC, Trace, BL, n=60, 127 | 0 | 0
  UWBC, 1+, BL, n=60, 127 | 1 | 6
  UWBC, 2+, BL, n=60, 127 | 0 | 1
  UWBC, 3+, BL, n=60, 127 | 1 | 0
  UWBC, Neg, Week 52/WD, n=56, 122 | 55 | 108
  UWBC, Trace, Week 52/WD, n=56, 122 | 0 | 0
  UWBC, 1+, Week 52/WD, n=56, 122 | 1 | 11
  UWBC, 2+, Week 52/WD, n=56, 122 | 0 | 3
  UWBC, 3+, Week 52/WD, n=56, 122 | 0 | 0

7. Secondary Outcome: Change From Baseline in 24-hour Urinary Cortisol Excretion at Weeks 24 and 52/Withdrawal (WD)
Description: 24-hour urinary cortisol excretion was calculated by multiplying the total volume of urine by the concentration of urinary cortisol. Cortisol is a hormone released from the adrenal gland that helps in fat, protein, and carbohydrate metabolism. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Week 0), Week 24, and Week 52/Withdrawal (WD)
Population: The Urine Cortisol Population: all participants in the ITT Population for whom a urine sample was obtained and whose urine sample was not considered to have confounding factors that could affect the interpretation of the results. Only those participants with post-Baseline data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles (nmol)/24 hours
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 25 | 43
Nanomoles (nmol)/24 hours
  Week 24, n=25, 43 | 1.0627 (76.135) | 0.8160 (55.926)
  Week 52/WD, n=24, 41 | 0.8862 (37.078) | 0.8593 (52.770)

8. Secondary Outcome: Change From Baseline in Blood Pressure at Weeks 4, 8, 12, 16, 24, 32, 40, and 52; Week 24/WD; and Week 52/WD
Description: Blood pressure measurement included systolic blood pressure (SBP) and diastolic blood pressure (DBP) at Weeks 4, 8, 12, 16, 24, 32, 40, and 52; Week 24/WD; and Week 52/WD. Blood pressure was measured in a sitting position after a participant was kept at rest for at least 5 minutes. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Week 0), Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 52, Week 24/WD, and Week 52/WD
Population: ITT Population. Only those participants with post-Baseline data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 58 | 125
Millimeters of Mercury (mmHg)
  SBP, Week 4, n=58, 124 | 4.3 (12.05) | 1.2 (12.47)
  SPB, Week 8, n=58, 123 | 2.5 (11.97) | 0.4 (13.33)
  SPB, Week 12, n=57, 119 | 2.7 (14.88) | 1.2 (14.00)
  SBP, Week 16, n=57, 116 | 1.2 (12.94) | 0.9 (14.18)
  SBP, Week 24, n=53, 115 | -0.3 (13.20) | -1.3 (14.63)
  SBP, Week 32, n=53, 112 | -1.8 (12.77) | -5.0 (14.76)
  SBP, Week 40, n=50, 107 | -3.0 (13.65) | -3.9 (14.06)
  SBP, Week 52, n=49, 106 | 3.7 (15.43) | 0.7 (15.16)
  SBP, Week 24/WD, n=56, 125 | -0.9 (13.73) | -1.1 (14.48)
  SBP, Week 52/WD, n=56, 123 | 2.4 (15.72) | 1.1 (15.82)
  DBP, Week 4, n=58, 124 | 3.3 (9.07) | 0.9 (10.13)
  DBP, Week 8, n=58, 123 | 0.1 (8.48) | 1.0 (9.55)
  DBP, Week 12, n=57, 119 | 0.7 (8.09) | 0.8 (10.76)
  DBP, Week 16, n=57, 116 | 0.4 (9.69) | 0.7 (10.76)
  DBP, Week 24, n=53, 115 | 0.3 (9.30) | -1.1 (11.71)
  DBP, Week 32, n=53, 112 | -1.6 (8.50) | -1.6 (11.23)
  DBP, Week 40, n=50, 107 | -1.6 (8.89) | -0.3 (11.08)
  DBP, Week 52, n=49, 106 | 1.2 (12.43) | 0.8 (10.77)
  DBP, Week 24/WD, n=56, 125 | 0.2 (9.34) | -1.2 (11.42)
  DBP, Week 52/WD, n=56, 123 | 0.8 (11.97) | 0.7 (11.29)

9. Secondary Outcome: Change From Baseline in Heart Rate (HR) at Weeks 4, 8, 12, 16, 24, 32, 40, and 52; Week 24/WD; and Week 52/WD
Description: Heart rate was measured in a sitting position after a participant was kept at rest for at least 5 minutes at assessment time points (Weeks 4, 8, 12, 16, 24, 32, 40, and 52; Week 24/WD; and Week 52/WD). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Week 0), Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 52, Week 24/WD, Week 52/WD
Population: ITT Population. Only those participants with post-Baseline data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats/Minute
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 58 | 125
Beats/Minute
  HR, Week 4, n=58, 124 | 0.2 (9.84) | -0.3 (11.04)
  HR, Week 8, n=58, 123 | -0.2 (11.41) | 0.3 (12.06)
  HR, Week 12, n=57, 119 | -1.6 (9.37) | -0.1 (11.27)
  HR, Week 16, n=57, 116 | 0.7 (9.50) | 1.5 (12.58)
  HR, Week 24, n=53, 115 | -0.7 (10.69) | -1.1 (11.53)
  HR, Week 32, n=53, 112 | -0.5 (9.23) | 0.1 (10.30)
  HR, Week 40, n=50, 107 | 1.7 (9.66) | -0.3 (11.59)
  HR, Week 52, n=49, 106 | 1.9 (9.32) | 1.1 (12.12)
  HR, Week 24/WD, n=56, 125 | -1.1 (11.03) | -0.7 (11.43)
  HR, Week 52/WD, n=56, 123 | 1.8 (10.62) | 2.0 (12.71)

10. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was recorded in a supine position after the participant was kept at rest in this position for at least 5 minutes at assessment time points (Week 12, Week 24, and Week52). Data are presented for clinically significant (CS) as well as not clinically significant (NCS) abnormal findings. Any abnormal ECG, including those that worsen from baseline, and clinically significant as assessed by the investigator were recorded as CS.
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Number analyzed (Participants) | 60 | 127
Participants
  BL, CS, n=60, 127 | 0 | 0
  BL, NCS, n=60, 127 | 19 | 43
  Week 12, CS, n=57, 119 | 0 | 1
  Week 12, NCS, n=57, 119 | 17 | 37
  Week 24, CS, n=54, 115 | 0 | 0
  Week 24, NCS, n=54, 115 | 17 | 33
  Week 52, CS, n=49, 106 | 1 | 1
  Week 52, NCS, n=49, 106 | 14 | 35

ADVERSE EVENTS:
Arm/Group | FF/VI 100/25 µg | FF/VI 200/25 µg
Serious Adverse Events (participants affected / at risk) | 10/60 | 23/127
Other Adverse Events (participants affected / at risk) | 36/60 | 93/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg (N=60) | FF/VI 200/25 µg (N=127)
Pneumonia (Infections and infestations) | 3 | 8
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Age-related macular degeneration (Eye disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg (N=60) | FF/VI 200/25 µg (N=127)
Nasopharyngitis (Infections and infestations) | 18 | 54
Bronchitis (Infections and infestations) | 5 | 8
Pharyngitis (Infections and infestations) | 4 | 7
Oral candidiasis (Infections and infestations) | 0 | 10
Pneumonia (Infections and infestations) | 1 | 8
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 13
Eczema (Skin and subcutaneous tissue disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.